CLINICAL TRIAL: NCT01480193
Title: Preliminary Clinical Trial of an Integrative Therapy With Severe Tinnitus
Brief Title: New Therapy for Patients With Severe Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00030594; 1R21DC011643-01 (NIH)
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-01

CONDITIONS: Tinnitus
Keywords: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: This pilot trial will employ a randomized controlled design in a 3:1 allocation series to gain experience with the experimental intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data management and analysis will be provided by blinded personnel.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sound Based and Educational Therapies (Active Comparator): The SBE program will consist of two hour-long individual counseling and sound therapy sessions based on the Department of Veterans Affairs Progressive Audiologic Tinnitus Management approach. SBE treatment incorporates the use of education, counseling, increased relaxation and decreased stress, along with the integration of sound therapy to better manage the impact of tinnitus.
  Interventions: Other: Sound Based and Educational Therapies
- Integrative Medicine Therapies and SBE (Experimental): 2 Sound Based and Educational Sessions 3 Cognitive Based Therapy Sessions 9 Telephonic Health Coaching Sessions 5 Acupuncture Sessions Group-Based 8 week Mindfulness Based Stress Reduction
  Interventions: Other: Sound Based and Educational Therapies; Other: Integrative Medicine Therapies and Sound Based Education Therapies

INTERVENTIONS:
Other: Sound Based and Educational Therapies — The SBE program will consist of two hour-long individual counseling and sound therapy sessions based on the Department of Veterans Affairs Progressive Audiologic Tinnitus Management approach. SBE treatment incorporates the use of education, counseling, increased relaxation and decreased stress, along with the integration of sound therapy to better manage the impact of tinnitus.
Other: Integrative Medicine Therapies and Sound Based Education Therapies — 3 Cognitive Based Therapy Sessions, 9 Telephonic Health Coaching Sessions, 5 Acupuncture Sessions, and Group-Based 8 week Mindfulness Based Stress Reduction Provided synergistically through an integrative medicine paradigm
  Arms: Integrative Medicine Therapies and SBE

SUMMARY:
Tinnitus is a common problem for which there is no universally effective treatment. The best available estimates indicate that 10 - 15% of adults report having tinnitus symptoms, but only 20% of those who report tinnitus suffer from it and subsequently seek treatment. Only formally reported by the U.S. Department of Veterans Affairs (VA), the economic impact of tinnitus is thought to be substantial. The VA reported in 2004 that 289,159 veterans received a disability award for their tinnitus amounting to a total annual compensation amount of over $345.5 million. Individuals with persistent severe tinnitus are unable to habituate to the tinnitus sound that most likely originates in the central auditory system (CAS) in response to peripheral injury. In a widely referenced study, it has been hypothesized that lack of habituation is secondary to abnormal processing of sensory information. Specifically, processing by the limbic system and autonomic nervous system is apparently abnormal in patients with increased levels of cortical arousal and inadequate coping mechanisms. In otolaryngology and audiology clinics, 'sound-based and educational therapies' (SBE) are the focus of most current therapies, and utilize enhanced sound input to the CAS. While SBE treatments may well provide a starting point for tinnitus treatment, additional treatment options are necessary particularly for those with significant non-auditory aspects of tinnitus (e.g., anxiety, depression, interference with daily life) as well as for those who do not experience significant improvement with SBE. Furthermore, commonly used forms of SBE [e.g.,Tinnitus Retraining Therapy (TRT)] can require over a year to become effective and may not be used in patients with hearing that is too poor to be modified by sound input. Based on prevalence data from tinnitus sufferers who seek treatment and the known percentage who do not respond to commonly used therapies, we estimate that 1.2 million individuals are not able to benefit at all from current, widely used treatment strategies. A new strategy to augment those currently used could empower patients to exert control over their tinnitus symptoms without the use of medications, expensive devices such as the Neuromonics device, or extended programs such as TRT. An alternative strategy may be useful both for patients who are not candidates for SBE and for those who respond poorly. An Integrative Medicine approach provides a likely solution. To date, there has been no systematic study of the benefits of an Integrative Medicine approach for severe tinnitus, particularly for non-auditory aspects of tinnitus symptoms. The goal of the proposed pilot study is to assess the feasibility of studying an integrative medicine approach in a subsequent large clinical trial which targets treatment of the non-auditory aspects of tinnitus suffering. Specifically, we wish to gain experience using the intervention in a randomized clinical trial when adding it to current commonly applied SBE therapies, compared with SBE alone. We also plan to assess patient satisfaction with the intervention, and obtain preliminary clinical efficacy data. If evaluating this intervention in an RCT appears feasible, this approach will be applied to a larger trial patient population in future studies to hypothesis test its efficacy and the durability of the potential effect. Our eventual goal is to develop a streamlined approach that individualizes tinnitus treatment based on symptoms and patient characteristics, and that can be widely applied in general medical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Debilitating tinnitus, defined by score on the Tinnitus Hearing Inventory > 38;
2. Participation not ruled out by baseline medical exam (see below);
3. Age 18 or older (no upper age limit);
4. No acute systemic illness requiring frequent treatment such as chemotherapy, dialysis, and no such treatment in the past 3 months,
5. Able to speak, read and write in English,
6. Willingness to participate fully in either treatment arm when randomized,
7. Not currently enrolled in another clinical trial or taking an experimental
8. No previous experience with either Sound Based and Educational (SBE) therapies as applied in this study or an Integrated Medicine approach specifically for the treatment of tinnitus symptoms; and
9. Adequate hearing to allow participation in the SBE treatment program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing the integrative medicine intervention in an RCT | baseline, 6 months post-baseline
  enrollment, retention, and patient feedback

SECONDARY OUTCOMES:
patient satisfaction | 6 months post-baseline
  Likert scales assessing patient perceptions of the integrative intervention

OTHER OUTCOMES:
Tinnitus-related dysfunction | baseline, 6 months post-baseline, 9 mos post baseline
  Tinnitus Handicap Questionnaire (THI) is a patient-reported survey that indicates dysfunction from tinnitus

CONTACTS AND LOCATIONS:
Overall Officials: Debara Tucci, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States